CLINICAL TRIAL: NCT01690650
Title: Oxygenation of the Neonatal Brain - a Study Using the INVOS Oximeter
Brief Title: Neonatal Cerebral Oxygenation After Exposure to Oxygen Evaluated With the INVOS Oximeter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: The Ludvig & Sara Elsass Foundation (Unknown)
Responsible Party: Principal Investigator, Line Carøe Sørensen, MD, PH.D., Copenhagen University Hospital, Hvidovre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Oxygen - HH 527
Record Dates: First submitted 2011-06-20; First posted 2012-09-24 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Response to Hyperoxia
Keywords: Preterm; Newborn; Neonate; Cerebral oxygenation; Oxygen
MeSH Terms: conditions — Premature Birth | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxygen + Cerebral NIRS (Experimental): Induced changes in oxygen supply (100% vs. room air). Continuously monitoring of cerebral oxygen saturation.
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — Oxygen exposure (100% oxygen) for 5 minutes, then 25 minutes with room air. Repeated twice. Continuously monitoring of the cerebral oxygen saturation (NIRS).5 replacements of sensor for reproducibility.

SUMMARY:
* Due to the increased risk of brain damage, continuous monitoring of the cerebral oxygenation is interesting. The investigators will evaluate the capability of the INVOS Oximeter to detect induced changes in the cerebral regional saturation.
* The purpose of the study is to investigate our hypothesis that cerebral vasoconstriction after oxygen exposure is prolonged in preterm infants compared to term infants.

DETAILED DESCRIPTION:
Preterm infants are at increased risk of brain damage compared with term infants, and cerebral hypoxia is considered to have an important role. The preterm infants are at increased risk of respiratory distress, episodes with low oxygenation, mechanical ventilation, risk of hypocapnia and labile or low blood pressure. These conditions can affect the microcirculation and hence the oxygenation of the brain. Hyperoxia is also a point of interest, since high levels of oxygen can cause vasoconstriction.

The investigators will examine the normal physiological cerebral response to exposure of oxygen in a group of preterm infants with a gestational age (GA) of 32-37 weeks and a group of term infants.

The investigators will do dynamic research with continuously monitoring of the cerebral oxygenation using the INVOS® Cerebral/Somatic Oximeter (Near InfraRed Spectroscopy (NIRS)). Reproducibility is examined by repeated measurements.

There will be no follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with a gestational age of 32-40 weeks
* Clinically stable
* +/- CPAP with a oxygen limit below 30%
* Parental consent

Exclusion Criteria:

* Severe birth asphyxia
* Prohibition of oxygen exposure

Ages: 1 Hour to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Changes from baseline of cerebral oxygen saturation after oxygen exposure. | Measurements will take between 30 minutes and 3 hours depending of situation. Measurements within the first 4 weeks of life. No follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ole Pryds, Professor, Principal Investigator — Department of Paediatrics, Copenhagen University Hospital, Hvidovre
Locations (1):
- Department of Paediatrics, Copenhagen University Hospital; Hvidovre, Hvidovre, Denmark